CLINICAL TRIAL: NCT01637727
Title: Long Term Effects of Gestational Diabetes Mellitus in a Population of Parous Women
Acronym: GDM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: GDM.CTIL; GDM.CTIL; GDMLTE.10
Record Dates: First submitted 2012-06-24; First posted 2012-07-11 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Long term effects of gestational diabetes mellitus in a population of parous women; Gestational diabetes mellitus- GDM is defined as glucose intolerance diagnosed during pregnancy and not present shortly after birth
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: the women will undergo a physical examination which will include measurements of blood pressure, height, weight and waist circumference.Blood samples will be obtained for evaluation of fasting glucose level, HbA1c, lipid profile and kidney functions.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GDM1: The study group will include women who gave birth in Shaare Zedek Medical Center between the years 2000 and 2010. Women with a GDM history will be identified based on the gestational diabetes clinic files. Women without a history of GDM who will be the control group will be identified from the Shaare Zedek Medical Center birth registration records.
- GDM: The study group will include women who gave birth in Shaare Zedek Medical Center between the years 2000 and 2010. Women with a GDM history will be identified based on the gestational diabetes clinic files. Women without a history of GDM who will be the control group will be identified from the Shaare Zedek Medical Center birth registration records.

SUMMARY:
The primary goal of this proposed research deals with estimating the risk of developing type 2 diabetes and metabolic syndrome in women with a history of GDM compared to women without a history of GDM. In addition, this study will attempt to evaluate the effect of parity on the late appearance of type 2 diabetes and metabolic syndrome in this unique population.

ELIGIBILITY:
Inclusion Criteria:

* The study group will include women who gave birth in Shaare Zedek Medical Center between the years 2000 and 2010.
* Women with a GDM history will be identified based on the gestational diabetes clinic files.
* Women without a history of GDM who will be the control group will be identified from the Shaare Zedek Medical Center birth registration records

Exclusion Criteria:

* We established the following exclusion criteria:

  * women who are diagnosed with metabolic syndrome before pregnancy or have type 1 or type 2 diabetes, and
  * women with severe chronic diseases.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The proposed research format is: a case control study using a historical cohort of women diagnosed with GDM. The study group will include women who gave birth in Shaare Zedek Medical Center between the years 2000 and 2010. Women with a GDM history will be identified based on the gestational diabetes clinic files. Women without a history of GDM who will be the control group will be identified from the Shaare Zedek Medical Center birth registration records
Sampling Method: Non-Probability Sample
Enrollment: 324 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Long term effects of gestational diabetes mellitus in a population of parous women | 24-32 months
  The primary goal of this proposed research deals with estimating the risk of developing type 2 diabetes and metabolic syndrome in women with a history of GDM compared to women without a history of GDM

SECONDARY OUTCOMES:
Long term effects of gestational diabetes mellitus in a population of parous women | 24-32 months.
  In addition, this study will attempt to evaluate the effect of parity on the late appearance of type 2 diabetes and metabolic syndrome in this unique population.

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Samueloff, Prof, Principal Investigator — Shaare Zedek Medical Center; Sorina Grissaro Granovsky, Dr, Study Chair — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel, Israel